CLINICAL TRIAL: NCT06744244
Title: Olfactory Memory in Infants With Signs of Asphyxia: An Early Indicator of Neurodevelopmental Outcomes
Brief Title: Olfactory Testing in Perinatal Asphyxia: Enhancing Risk Assessment
Acronym: MEMOBRAIN
Status: Recruiting | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Serafina Perrone, Professor, University of Parma
Other Study IDs: 27408
Record Dates: First submitted 2024-12-06; First posted 2024-12-20 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Mild Birth Asphyxia; Moderate Birth Asphyxia
Keywords: Perinatal Asphyxia; Hypoxic-Ischemic Encephalopathy; Biomarkers; Olfactory Function
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Heart Rate; Respiratory Rate; Oxygen Saturation; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild Birth Asphyxia: Term newborns (37-41 weeks of gestational age) with signs of moderate asphyxia at birth (cord pH < 7.10 and/or BE > -12), with mild asphyxia at birth.
  Interventions: Diagnostic Test: Olfactory Testing; Diagnostic Test: Heart rate (HR), Heart Rate Variability (HRV), Respiratory Rate (RR), peripheral oxygen saturation (SpO2); Diagnostic Test: Video-EEG; Diagnostic Test: fMRI; Diagnostic Test: Neurodevelopment assessment
- Moderate - Severe Birth Asphyxia: Term newborns (37-41 weeks of gestational age) with signs of moderate asphyxia at birth (cord pH < 7.10 and/or BE > -12) with moderate asphyxia at birth, at risk of developing hypoxic-ischemic encephalopathy, who don't need hypothermia treatment and with severe asphyxia at birth, at risk of developing hypoxic-ischemic encephalopathy who don't need hypothermia treatment.
  Interventions: Diagnostic Test: Olfactory Testing; Diagnostic Test: Heart rate (HR), Heart Rate Variability (HRV), Respiratory Rate (RR), peripheral oxygen saturation (SpO2); Diagnostic Test: Video-EEG; Diagnostic Test: fMRI; Diagnostic Test: Neurodevelopment assessment

INTERVENTIONS:
Diagnostic Test: Olfactory Testing — Olfactory Test: Odor stimuli will be administered using a custom-designed olfactometer, developed by engineers specifically for this study. The olfactometer will release different odorants (maternal breast milk, vanilla essential oil, rose essential oil, and water as a control) in a controlled way. Each odor will be presented between 6 and 72 hours of life for 10 seconds (On), followed by a 50-second pause (Off) for a total of 15 cycles (On-Off). A new odor will be presented 5 minutes after the previous one. The first olfactory test will be conducted during the Video-EEG recording, and the second one will take place during the fMRI acquisition.
Diagnostic Test: Heart rate (HR), Heart Rate Variability (HRV), Respiratory Rate (RR), peripheral oxygen saturation (SpO2) — Simultaneously with the presentation of odors, heart rate (HR), heart rate variability (HRV), respiratory rate (RR), and peripheral oxygen saturation (SpO2) will be monitored and recorded. The onset of the odor will be recorded using a manual timer.
Diagnostic Test: Video-EEG — The infant's Video-EEG, as per guidelines following perinatal asphyxia, will be recorded for approximately 2 hours, including the period preceding odor administration (baseline).
Diagnostic Test: fMRI — Newborns will undergo an fMRI, as part of routine clinical practice, to identify any brain injury, its extent, and the structures involved. The use of a custom-built fMRI compatible olfactometer will facilitate these studies.
Diagnostic Test: Neurodevelopment assessment — Between 12 and 18 months, the infants will undergo neurodevelopmental follow-up, during which the Bayley III assessment will be administered to evaluate any potential neurocognitive deficits.

SUMMARY:
Neonatal asphyxia remains a leading cause of neurodevelopmental disabilities despite advancements in perinatal care. Hypoxic-ischemic encephalopathy (HIE), a severe outcome of asphyxia, impacts 1-3 infants per 1,000 live births annually in industrialized nations, causing long-term neurological impairments such as cognitive dysfunction, motor deficits, and sensory impairments. Early identification of at-risk newborns is critical to initiate timely interventions and improve outcomes.

Olfactory perception, crucial for newborns' adaptation to extrauterine life, involves odor identification and memory. Odor perception is known to be impaired in adults with neurological disorders and in animal models of brain injury. However, no clinical studies have assessed olfactory function in newborns with signs of asphyxia. Olfactory memory, which can be evaluated through habituation to repeated odors, may provide insights into early brain function.

This study aims to evaluate whether olfactory memory can serve as an early marker of neurodevelopmental outcomes in newborns with signs of asphyxia. By assessing physiological, behavioral, and neurological responses to olfactory stimuli, the study seeks to explore the differences between infants with mild asphyxia and those with moderate-to-severe asphyxia.

DETAILED DESCRIPTION:
Neonatal asphyxia is the leading cause of neurodevelopmental disability. Despite recent advances in perinatal medicine, which have improved associated mortality, the neurological outcomes of hypoxic-ischemic events in newborns remain significant. The incidence of neonatal asphyxia is estimated to be 1.5 per 100 live births per year in industrialized countries with advanced obstetric-neonatal care. Between 1 and 3 infants per 1,000 live births suffer from severe neurological impairment due to perinatal asphyxia, developing hypoxic-ischemic encephalopathy.

Early identification of newborns with signs of asphyxia who are at high risk for hypoxic-ischemic encephalopathy and brain damage can improve outcomes by enabling the early initiation of rehabilitative interventions. Hypoxic-ischemic injury often results in impairments in audiovisual perception, cerebral palsy, cognitive dysfunction, memory difficulties, and other neurological sequelae.

Olfactory perception (the sense of smell) is one of the most important sensory functions in humans. In newborns, the sense of smell plays a crucial role, allowing them to perceive maternal odors and breast milk, guiding them in adapting to their environment and completing the physiological transition from intrauterine to extrauterine life. Olfactory neurosensory function involves several abilities, particularly odor identification and memory. Olfactory perception is also linked to olfactory memory, which can be tested as a habituation response. Olfactory memory is defined as the recollection of odorants. In recent studies, exposure to pleasant odors, such as breast milk or vanilla, has been shown to reduce perceived pain during invasive procedures in healthy full-term newborns. Olfactory stimuli can generate various physiological changes, regulating heart and respiratory rates, as well as triggering motor responses that guide head movements and initiate orofacial responses.

Some studies have shown that brain injury impairs odor perception: smell is altered in several neurological conditions, including both neurodevelopmental and neurodegenerative disorders. In Alzheimer (AD), Parkinson disease (PD) and in stroke, several cortical and subcortical areas directly involved in olfactory function are damaged or show signs of atrophy, including the olfactory bulb (OB), primary olfactory cortex (POC), hippocampus, orbitofrontal cortex (OFC), amygdala, and olfactory tract. Moreover, reduced odor detection early in life, along with anatomical and functional alterations in olfactory and higher-order cortical networks, has been reported in neurodevelopmental disorders such as Autistic Spectrum Disorder (ASD) and Attention Deficit / Hyperactivity Disorder (ADHD).

Olfactory dysfunction has also been studied and demonstrated in animal models through the induction of brain damage in rabbits. So far, no study has evaluated olfactory function in the clinical setting of brain injury due to neonatal asphyxia.

In cases of perinatal asphyxia, early identification of hypoxic-ischemic encephalopathy is achieved through continuous video-electroencephalographic monitoring, which is currently considered the gold standard for evaluating brain functions and detecting subclinical seizures. Although EEG does not directly assess olfactory function, certain electroencephalographic alterations may suggest impairment in brain regions involved in olfactory perception (piriform cortex, insular cortex, and amygdala).There are numerous studies in the literature that adopt various methods of olfactory testing in healthy newborns, but no validated tool or test exists to evaluate olfactory memory in newborns.

This study aims to assess olfactory function in newborns exhibiting signs of asphyxia at birth and to investigate whether infants with mild asphyxia differ from those with moderate to severe asphyxia.

The hypotheses of this study is that olfactory stimulation with odors such as rose, vanilla, and breast milk induces changes in heart rate, respiratory rate, peripheral oxygen saturation, EEG activity, and neuroimaging measures in asphyxiated newborns. These changes also occur following repeated olfactory stimuli. Olfactory memory, or habituation to odors, is delayed or absent in newborns with moderate-severe asphyxia.

ELIGIBILITY:
Inclusion Criteria:

* Term newborns (37-41 weeks of gestational age) with signs of asphyxia at birth (cord pH < 7.10 and/or BE > -12).
* Maternal age > 18 years.
* No medication use during pregnancy (e.g., antipsychotics, antidepressants, sedatives, anticonvulsants, anxiolytics).
* Absence of maternal infections.
* Apgar score < 5 at 10 minutes of life.
* Newborns with mild asphyxia at birth.
* Newborns with moderate asphyxia at birth, at risk of developing hypoxic-ischemic encephalopathy, who don't need hypothermia treatment.
* Newborns with severe asphyxia at birth, at risk of developing hypoxic-ischemic encephalopathy who don't need hypothermia treatment.

Exclusion Criteria:

* Post-term infants (gestational age > 42 weeks).
* Preterm infants (gestational age < 37 weeks).
* Infants with genetic syndromes or congenital anomalies.
* Infants from mothers using drugs of abuse.
* Infants with scalp injuries or lesions.
* Infants with microcephaly.
* Infants who underwent therapeutic hypothermia.

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns with signs of mild asphyxia and newborns with signs of moderate-severe asphyxia at high risk for hypoxic-ischemic encephalopathy and brain damage.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Autonomic Responses to Olfactory Stimulation in Asphyxiated Newborns. | during the Olfactory Testing
  Heart Rate (HR) and Heart Rate Variability (HRV) will be continuously monitored via electrocardiography throughout the procedure and compared between the two groups. Data will be analyzed using software such as Kubios.
  For HRV, the following metrics will be extracted:
  SDNN (Standard Deviation of NN Intervals): Reflects overall HRV. RMSSD (Root Mean Square of Successive Differences): Reflects parasympathetic (vagal) activity.
  LF Power (Low-Frequency): Reflects both sympathetic and parasympathetic activity (0.04 - 0.15 Hz).
  HF Power (High-Frequency): Primarily reflects parasympathetic activity (0.15 - 0.4 Hz).
  LF/HF Ratio: Assesses the balance between sympathetic and parasympathetic activity, with a higher ratio indicating sympathetic dominance.
Breathing patterns in Asphyxiated Newborns. | during the Olfactory Testing
  Variations in breathing patterns are assessed by the pulse oximeter that operates on the principle of light absorption, emitting red and infrared light through the skin. A photodetector measures the light absorbed by the blood, with oxygenated hemoglobin absorbing more infrared light and deoxygenated hemoglobin absorbing more red light. The ratio of light absorption at these wavelengths is used to estimate the percentage of oxygenated hemoglobin (Peripheral Oxygen Saturation - SpO2), displayed as a percentage on the device's screen. This metric provides insight into oxygenation levels in the bloodstream, which may improve due to enhanced respiratory efficiency triggered by olfactory exposure. The pulse oximeter also features a respiratory rate (RR) measurement, estimating RR by detecting changes in blood flow or pulse linked to breathing patterns.
Cerebral functioning in Asphyxiated Newborns. | Within 6 to 72 hours of life
  Amplitude EEG (aEEG) provides a continuous, real-time overview of cerebral function by measuring the brain's electrical activity. In the context of perinatal asphyxia, aEEG is used to detect abnormal brain patterns, such as reduced or absent brain activity. These patterns are reflected in the amplitude of the signal (measured in microvolts), which can indicate the severity of brain injury and help clinicians assess the extent of neurological damage.
Changes in olfactory evoked potentials (EOPs) in Asphyxiated Newborns. | during the Olfactory Testing
  The analysis of EOPs in response to olfactory stimuli, such as rose, vanilla, and breast milk, will be conducted using dedicated software like EEGLAB and ERPLAB (MATLAB). The analysis parameters for EOPs will include latency, amplitude, wave components, spatial distribution, duration, topography and localization, as well as habituation and adaptation. These parameters will be compared between the two groups.
Spectral analysis of brain oscillatory rhythms to monitor changes in global brain activity. | Within 6 to 72 hours of life
  Brain activity will be continuously monitored with electroencephalography (EEG) throughout the procedure using a 12-channel system and oscillatory activity across brain rhythm bands (Delta: 0.5 - 4 Hz, Theta: 4 - 8 Hz, Alpha: 8 - 12 Hz, Beta: 12 - 30 Hz, Gamma: 30 - 100 Hz) will be analyzed with dedicated software such as EEGLAB (MATLAB) in both groups.
Changes in behavioral responsens to Olfactory Stimulation in Asphyxiated Newborns. | Within 6 to 72 hours of life
  Facial expressions obtained from video-recordings will be assessed by two neonatologists, who will be blinded to the odor used to obtain insight into changes in behavioral responsens.
  A score will be assigned on a scale of 0 to 100 (0 = extremely disgusted; 100 = extremely pleased).
  The neonatologists will view the video as many times as necessary to ensure the highest accuracy inscoring. The videos will be destroyed after 5 years.
Highlight a different activation within brain areas involved in olfactory perception, memory, and learning through fMRI. | Within 6 to 72 hours of life
  Data from functional magnetic resonance imaging (fMRI) will be analyzed to compare the activation of regions of interest (ROIs), especially in regions such as the olfactory bulb, entorhinal cortex, hippocampus, and amygdala, between the two groups of patients during the execution of olfactory test. The parameters that will be evalueted and compared between the two groups will be: BOLD Signal (Blood Oxygenation Level Dependent), Activation Intensity (Signal Strength), Peak Activation, Time Course of Activation, Functional Connectivity and Effect Size.

SECONDARY OUTCOMES:
Neurodevelopmental follow-up | Between 12 and 18 months
  The Bayley III assessment will be administered in both groups. It provides a comprehensive overview of a child's cognitive, motor, and socio-emotional abilities. The measures obtained from the Bayley-III include cognitive, motor, language, social-emotional and adaptive behavior scales. Scores from the different scales are converted into standard scores (mean of 100, standard deviation of 15), which help compare the child to the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Serafina Perrone, MD, PhD, Principal Investigator — Università di Parma
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, Italy

REFERENCES:
- [Background] Chavez-Valdez R, Miller S, Spahic H, Vaidya D, Parkinson C, Dietrick B, Brooks S, Gerner GJ, Tekes A, Graham EM, Northington FJ, Everett AD. Therapeutic Hypothermia Modulates the Relationships Between Indicators of Severity of Neonatal Hypoxic Ischemic Encephalopathy and Serum Biomarkers. Front Neurol. 2021 Nov 2;12:748150. doi: 10.3389/fneur.2021.748150. eCollection 2021. PMID 34795631
- [Background] Finder M, Boylan GB, Twomey D, Ahearne C, Murray DM, Hallberg B. Two-Year Neurodevelopmental Outcomes After Mild Hypoxic Ischemic Encephalopathy in the Era of Therapeutic Hypothermia. JAMA Pediatr. 2020 Jan 1;174(1):48-55. doi: 10.1001/jamapediatrics.2019.4011. PMID 31710357
- [Background] Ambalavanan N, Shankaran S, Laptook AR, Carper BA, Das A, Carlo WA, Cotten CM, Duncan AF, Higgins RD; EUNICE KENNEDY SHRIVER NICHD NEONATAL RESEARCH NETWORK. Early Determination of Prognosis in Neonatal Moderate or Severe Hypoxic-Ischemic Encephalopathy. Pediatrics. 2021 Jun;147(6):e2020048678. doi: 10.1542/peds.2020-048678. Epub 2021 May 13. PMID 33986149
- [Background] Disdier C, Stonestreet BS. Hypoxic-ischemic-related cerebrovascular changes and potential therapeutic strategies in the neonatal brain. J Neurosci Res. 2020 Jul;98(7):1468-1484. doi: 10.1002/jnr.24590. Epub 2020 Feb 14. PMID 32060970
- [Background] Drobyshevsky A, Robinson AM, Derrick M, Wyrwicz AM, Ji X, Englof I, Tan S. Sensory deficits and olfactory system injury detected by novel application of MEMRI in newborn rabbit after antenatal hypoxia-ischemia. Neuroimage. 2006 Sep;32(3):1106-12. doi: 10.1016/j.neuroimage.2006.06.002. Epub 2006 Jul 24. PMID 16861007
- [Background] Juliano C, Sosunov S, Niatsetskaya Z, Isler JA, Utkina-Sosunova I, Jang I, Ratner V, Ten V. Mild intermittent hypoxemia in neonatal mice causes permanent neurofunctional deficit and white matter hypomyelination. Exp Neurol. 2015 Feb;264:33-42. doi: 10.1016/j.expneurol.2014.11.010. Epub 2014 Dec 2. PMID 25476492
- [Background] Schaal B, Saxton TK, Loos H, Soussignan R, Durand K. Olfaction scaffolds the developing human from neonate to adolescent and beyond. Philos Trans R Soc Lond B Biol Sci. 2020 Jun 8;375(1800):20190261. doi: 10.1098/rstb.2019.0261. Epub 2020 Apr 20. PMID 32306879
- [Background] Tristao RM, Lauand L, Costa KSF, Brant LA, Fernandes GM, Costa KN, Spilski J, Lachmann T. Olfactory sensory and perceptual evaluation in newborn infants: A systematic review. Dev Psychobiol. 2021 Nov;63(7):e22201. doi: 10.1002/dev.22201. PMID 34674234
- [Background] Chen X, Gao F, Lin C, Chen A, Deng J, Chen P, Lin M, Xie B, Liao Y, Gong C, Zheng X. mTOR-mediated autophagy in the hippocampus is involved in perioperative neurocognitive disorders in diabetic rats. CNS Neurosci Ther. 2022 Apr;28(4):540-553. doi: 10.1111/cns.13762. Epub 2021 Nov 16. PMID 34784444
- [Background] Lan HY, Yang L, Lin CH, Hsieh KH, Chang YC, Yin T. Breastmilk as a Multisensory Intervention for Relieving Pain during Newborn Screening Procedures: A Randomized Control Trial. Int J Environ Res Public Health. 2021 Dec 10;18(24):13023. doi: 10.3390/ijerph182413023. PMID 34948633
- [Background] Baudesson de Chanville A, Brevaut-Malaty V, Garbi A, Tosello B, Baumstarck K, Gire C. Analgesic Effect of Maternal Human Milk Odor on Premature Neonates: A Randomized Controlled Trial. J Hum Lact. 2017 May;33(2):300-308. doi: 10.1177/0890334417693225. Epub 2017 Mar 27. PMID 28346843
- [Background] Zhang S, Su F, Li J, Chen W. The Analgesic Effects of Maternal Milk Odor on Newborns: A Meta-Analysis. Breastfeed Med. 2018 Jun;13(5):327-334. doi: 10.1089/bfm.2017.0226. Epub 2018 May 7. PMID 29733222
- [Background] Doucet S, Soussignan R, Sagot P, Schaal B. The "smellscape" of mother's breast: effects of odor masking and selective unmasking on neonatal arousal, oral, and visual responses. Dev Psychobiol. 2007 Mar;49(2):129-38. doi: 10.1002/dev.20210. PMID 17299785
- [Background] Schaal B, Marlier L, Soussignan R. Responsiveness to the odour of amniotic fluid in the human neonate. Biol Neonate. 1995;67(6):397-406. doi: 10.1159/000244192. PMID 7578623
- [Background] Schaal B, Marlier L, Soussignan R. Olfactory function in the human fetus: evidence from selective neonatal responsiveness to the odor of amniotic fluid. Behav Neurosci. 1998 Dec;112(6):1438-49. doi: 10.1037//0735-7044.112.6.1438. PMID 9926826
- [Background] Schleidt M & Genzel C, The significance of mother's perfume for infants in the first weeks of their life. Ethology and Sociobiology. 1990; 11(3); 145-154. https://doi.org/10.1016/0162-3095(90)90007-S
- [Background] Varendi H, Christensson K, Porter RH, Winberg J. Soothing effect of amniotic fluid smell in newborn infants. Early Hum Dev. 1998 Apr 17;51(1):47-55. doi: 10.1016/s0378-3782(97)00082-0. PMID 9570031
- [Background] Soussignan R, Schaal B, Marlier L. Olfactory alliesthesia in human neonates: prandial state and stimulus familiarity modulate facial and autonomic responses to milk odors. Dev Psychobiol. 1999 Jul;35(1):3-14. doi: 10.1002/(sici)1098-2302(199907)35:13.0.co;2-f. PMID 10397891
- [Background] Soussignan R, Schaal B, Marlier L, Jiang T. Facial and autonomic responses to biological and artificial olfactory stimuli in human neonates: re-examining early hedonic discrimination of odors. Physiol Behav. 1997 Oct;62(4):745-58. doi: 10.1016/s0031-9384(97)00187-x. PMID 9284493
- [Background] Bersani I, Piersigilli F, Gazzolo D, Campi F, Savarese I, Dotta A, Tamborrino PP, Auriti C, Di Mambro C. Heart rate variability as possible marker of brain damage in neonates with hypoxic ischemic encephalopathy: a systematic review. Eur J Pediatr. 2021 May;180(5):1335-1345. doi: 10.1007/s00431-020-03882-3. Epub 2020 Nov 27. PMID 33245400
- [Background] Murray DM, Boylan GB, Ryan CA, Connolly S. Early EEG findings in hypoxic-ischemic encephalopathy predict outcomes at 2 years. Pediatrics. 2009 Sep;124(3):e459-67. doi: 10.1542/peds.2008-2190. Epub 2009 Aug 24. PMID 19706569
- [Background] Allegaert K, van de Velde M, van den Anker J. Neonatal clinical pharmacology. Paediatr Anaesth. 2014 Jan;24(1):30-8. doi: 10.1111/pan.12176. Epub 2013 Apr 26. PMID 23617305
- [Background] Boylan GB, Stevenson NJ, Vanhatalo S. Monitoring neonatal seizures. Semin Fetal Neonatal Med. 2013 Aug;18(4):202-8. doi: 10.1016/j.siny.2013.04.004. Epub 2013 May 24. PMID 23707519
- [Background] Shellhaas RA, Soaita AI, Clancy RR. Sensitivity of amplitude-integrated electroencephalography for neonatal seizure detection. Pediatrics. 2007 Oct;120(4):770-7. doi: 10.1542/peds.2007-0514. PMID 17908764
- [Background] Elshorbagy HH, Azab AA, Kamal NM, Barseem NF, Bassiouny MM, Elsayed MA, Elkhouly TH. Value of electroencephalographic monitoring in newborns with hypoxic-ischemic encephalopathy treated with hypothermia. J Pediatr Neurosci. 2016 Oct-Dec;11(4):309-315. doi: 10.4103/1817-1745.199467. PMID 28217152
- [Background] Cloherty, J. P., Eichenwald, E. C., Stark, A. R., & Hansen, A. R. (Eds.). (2016). Cloherty and Stark's Manual of Neonatal Care (8th ed.). Philadelphia, PA: Wolters Kluwer.